CLINICAL TRIAL: NCT00150475
Title: Contamination During Removal of Two Different Personal Protective Systems When Working Under Conditions Requiring Enhanced Respiratory and Contact Precautions
Brief Title: Contamination During Removal of Two Different Personal Protective Systems
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University (Other)
Collaborators: The Physicians' Services Incorporated Foundation (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Educational/Counseling/Training
Other Study IDs: PSI 04-58
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2005-09-08 (Estimated); Status verified 2005-09

CONDITIONS: Severe Acute Respiratory Syndrome
Keywords: Severe Acute Respiratory Syndrome
MeSH Terms: conditions — Severe Acute Respiratory Syndrome

INTERVENTIONS:
Procedure: Powered Air purifying respirator

SUMMARY:
Highly communicable and virulent diseases, the ongoing threat of emerging infectious diseases, and the prospect of bio-terrorism have become part of the new reality for health care workers. SARS transmission has occurred despite the use of droplet, contact, and airborne precautions. Potential explanations for some of the episodes of "through-precautions" transmission include the possibility of contamination during removal of protective clothing.

The recommended protective systems (PPS) for aerosol generating procedures set out by the US Center for Disease Control and Prevention (CDC) and the Ontario Ministry of Health and Long Term Care (MOHLTC) differ.

The failure of a PPS may be associated with significant consequences in terms of the morbidity and mortality of front-line health care workers. The purpose of this study is to determine if a difference exists between the rate of self-contamination due to deficiencies in contact precautions for individuals wearing either the CDC or MOHLTC recommended PPS.

Study participants will don one of the two recommended PPS, be "contaminated" with an indicator that becomes visible under ultraviolet light, and then assessed for contamination of clothing layers and skin after removal of the PPS. They will then repeat the procedure using the other PPS.

DETAILED DESCRIPTION:
Background: Highly communicable and virulent diseases such as severe acute respiratory syndrome (SARS) and "avian influenza", the ongoing threat of other emerging infectious diseases, and the prospect of bio-terrorism have become part of the new reality for health care workers (1). Recent experience with SARS has demonstrated that front-line health care professionals who perform or assist with aerosol generating procedures are at particularly increased risk of infection.

At present, no data exists addressing the question of self-contamination during the removal of personal protective systems used in a health care setting. The latest suggested donning and removal procedures have not been validated with respect to the issue of selfcontamination due to deficiencies in contact precautions.

The failure of a personal protective system or the donning and removal procedures for a personal protective system may be associated with significant consequences in terms of the morbidity and mortality of front-line health care workers. It is imperative that the rate of self-contamination for these two personal protective systems be assessed.

The purpose of this study is to determine if a difference exists between the rate of self-contamination due to deficiencies in contact precautions for individuals wearing either Personal Protective Equipment (PPE) or the Powered Air Purifying Respirator (PAPR).

This will be a prospective, randomized, controlled, crossover study.

Institutional Ethics Committee approval will be obtained for this study. Fifty participants will be required for the study. Participants will be recruited from the Department of Anesthesiology attending and resident staff, other physician groups requiring PAPR training, and the Department of Respiratory Therapy. Recruitment will occur in conjunction with annual training in the use of the PAPR. Individuals will be informed of the purpose and procedure of the study and written consent will be obtained. Individuals will be excluded if they refuse to provide written consent to participate in the study.

Participants will wear operating room scrub attire as their base clothing layer.

They will be randomized to don either the PAPR or PPE. They will then repeat the process using the other personal protective system immediately after the study protocol has been completed using the first personal protective system.

PPE will consist of an N95 respirator, goggles, face shield, bouffant hair cover, fluid resistant surgical gown, and fitted sterile gloves. Although the CDC has omitted a head covering as part of their PPE, the MOHLTC directives stipulate that a head covering must be worn when performing high-risk procedures in patients that require enhanced respiratory and contact precautions. A head covering (bouffant hair cover) will therefore form part of the PPE used in this study. The CDC recommendations state that goggles can be worn for eye protection. A face shield can be used in addition to the goggles but this is optional. The MOHLTC directives state that goggles and a face shield must be worn during high-risk procedures in patients that require enhanced respiratory and contact precautions. Goggles and a face shield will therefore form part of the PPE for this study. Therefore the donning and removal instructions for the PPE that will be used for this study will differ in sequence from those published by the CDC. The donning and removal procedures that will be used for this study more closely follow the sequence recommended by the MOHLTC and are indeed an enhanced version of those directives.

PAPR will consist of a body suit and shoe covers, PAPR hood and power unit, N95 respirator, goggles, face shield, bouffant hair cover, fluid resistant surgical gown, and fitted sterile gloves. The MOHLTC has stipulated the use of donning/removal coaches for the PAPR. Neither the CDC, the MOHLTC, nor our institution have stipulated the use of donning/removal coaches for the PPE. The intent of this study is to examine the protective systems. The donning and removal procedures that form part of the protective systems may either contribute to or minimize self-contamination rates and must be assessed under the actual conditions of use. In order to best simulate the actual conditions that health care workers will be subjected to and to best evaluate donning and removal procedures and practices we have also decided not to employ a donning/removal coach for the PPE. Accordingly, during donning and removal of PPE participants will be given standardized written instructions outlining the donning and removal procedure but will not be coached.

Participants will be given standardized written instructions and coached by a respiratory therapist during donning and removal of the PAPR. The standardized written instructions for donning and removal of both the PPE and PAPR are attached in Appendices A and B.

All participants will be timed and videotaped during the protective system donning procedure. Timing will commence when the participants are instructed to begin reading 3 their written donning instructions for PPE or when the dressing coach says "begin" for the PAPR. Timing will cease when the participants have completed donning the final item of the protective system being tested. Videotaping will occur in order to record and assist in the detection of any protective system donning procedure violations. A donning procedure violation will be defined as having occurred if the participants perform a donning maneuver out of sequence or touch a piece of protective equipment out of sequence. Participants will be "contaminated" using a solution of fluorescein (1ml of a 25% solution diluted in 100cc sterile water) in a standardized fashion. A Devilbiss atomizer (Model DV-15-RD, Sunrise Medical Products, Carlsbad, California, USA) will be used to apply 5ml of fluorescein solution to the their front face shield and torso. We have chosen these contamination sites in order to simulate areas that would most likely be contaminated by the large respiratory droplets aerosolized by a patient that is either coughing or reacting to intubation attempts or any other high-risk respiratory procedure.

The atomizer nozzle will be held at a distance of 30cm from the participants' face-shield and will be applied from their shoulder level. The spray stream will be directed at the participants' nose and then aimed inferiorly towards the their umbilicus in an upwards and downwards sweeping motion while keeping the atomizer oriented in the participants' mid-saggital plane. Application will occur until the atomizer reservoir is empty. During this application the participants' eyes will be closed. "Invisible" Detection Paste (Sirchie, 100 Hunter Place, Youngsville, NC) will be applied to the palmar aspects of the participants' hands and anterior and posterior forearm to the elbow. Although the paste is labeled "invisible detection paste" it becomes visible when viewed under ultraviolet (UV) light. 15ml of paste will be used. We have chosen to use detection paste on the forearms and gloves of the study participants as these are the areas most likely to come in contact with any patient requiring enhanced contact and respiratory precautions. Participants will be videotaped, photographed with a digital camera, and assessed with a UV lamp (Burton Medical Products Inc, 21100 Lassen Street, Chatsworth, CA. 91311 USA) following contamination to ensure that standardized contamination of their front face shield, torso, forearm, and palmar aspect of the gloved hands has been achieved.

Participants will then follow the standardized written removal procedures for the protective system that they are wearing. They will be timed and videotaped during the protective system removal procedure. Timing will commence when the participants are instructed to begin reading their written removal instructions for PPE or when the dressing coach says "begin" for the PAPR. Timing will be paused during assessments with the UV lamp. Timing will cease when the participants have completed removing the final item of the protective system being tested. Videotaping will occur in order to record and assist in the detection of any protective system removal procedure violations. A removal procedure violation will be defined as having occurred if the participants perform a removal maneuver out of sequence, touch a piece of protective equipment out 4 of sequence, or touch any part of their body other than a piece of protective equipment prior to performing final hand disinfection. Participants will be assessed with the UV lamp at specific intervals during the removal procedure in order to detect any visible contamination. Participants in PPE will be assessed with the UV lamp following removal of the outer PPE protective layer (outer fitted sterile gloves, fluid resistant surgical gown, and faceshield).

Final assessment will occur after removal of the inner PPE protective layer (N95 mask, goggles, bouffant hair cover, inner fitted sterile gloves). Participants in PAPR will be assessed using the UV lamp after removal of the outer PAPR protective layer (PAPR hood and power unit, outer fluid resistant surgical gown, outer boot covers, outer fitted sterile gloves). They will then be assessed after removal of the middle PAPR protective layer (body suit, middle sterile fitted gloves, boot covers).

Final assessment will occur after removal of the inner PAPR protective layer (N95 mask, goggles, bouffant hair cover, inner sterile fitted gloves). An evaluator blinded to the participants' protective system will perform final assessment.

All areas of the participants' base clothing layer and any exposed skin and hair will be inspected after removal of the final protective layer. This will include the participants' face. Contamination episodes will be counted and the contamination area will be calculated in cm2.

ELIGIBILITY:
Inclusion Criteria:Participants will be recruited from the Department of Anesthesiology attending and resident staff, other physician groups requiring PAPR training, and the Department of Respiratory Therapy.

-

Exclusion Criteria:Individuals will be excluded if they refuse to provide written consent to participate in the study

-

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2005-01; Study Completion 2005-05

PRIMARY OUTCOMES:
The primary endpoint of this study is the presence of any detected
base clothing layer, skin, or hair contamination.

SECONDARY OUTCOMES:
The secondary endpoints: 1) contamination episodes of any layer, and 2) protective
system donning and removal procedure violations

CONTACTS AND LOCATIONS:
Overall Officials: Jorge E. Zamora, MD, Principal Investigator — Queen's University
Locations (1):
- Kingston General Hospital, Kingston, Ontario, Canada